CLINICAL TRIAL: NCT07326254
Title: Determining the Effectiveness of Chewing Gums With Different Flavors in Reducing Procedural Pain and Fear in Children Aged 7 to 12
Brief Title: Effect of Chewing Different Flavor Gum on Procedural Pain and Fear
Acronym: Gum-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Emine Beyaz, Principal Investigator, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MusAl
Record Dates: First submitted 2025-11-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
Keywords: pain management; chewing gum; pediatric nursing; venipuncture; anxiety
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants were randomly assigned to three groups: control (no gum), sugared gum, and sugar-free gum (n = 48 each) . Randomization was performed using sealed opaque envelopes labeled with group codes. Each child selected one envelope in the presence of a parent. The nurse who performed the blood draw and the researcher responsible for data collection were blinded to group allocation. Complete participant blinding was not feasible due to the visible nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sugared Gum (Experimental): Participants start chewing sugared gum one minute before the procedure and continue chewing until the procedure is over.
  Interventions: Behavioral: Sugared Gum Chewing
- Sugar-Free Gum (Experimental): Participants start chewing sugared gum one minute before the procedure and continue chewing until the procedure is over.
  Interventions: Behavioral: Sugar-Free Gum Chewing
- Control (Placebo Comparator): This group did not receive any gum chewing intervention during the blood collection procedure. Standard procedures were followed. The parent was present with the child during the procedure.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Sugared Gum Chewing — Chewing sugared gum, which began one minute before the procedure, continued until the end of the blood collection. Sugared gum provided a sweet taste stimulus, while sugarless gum served as a non-sweet comparator. Children were continuously monitored to ensure safety and prevent aspiration, and children aged 7-12 were included in the study. No adverse events were reported during the study.
  Arms: Sugared Gum
Behavioral: Sugar-Free Gum Chewing — Participants began chewing sugarless gum one minute before the procedure began, until the blood sample was collected. The purpose of the chewing activity was to reduce pain and fear during the procedure. No other behavioral or pharmacological interventions were administered.
  Arms: Sugar-Free Gum
Other: Control — No active gum chewing intervention was performed during blood collection
  Arms: Control

SUMMARY:
Needle-related pain and anxiety present persistent challenges in pediatric clinical procedures. This study aims to investigate the effects of chewing sugared and sugar-free gum on pain, anxiety, and fear in children undergoing venipuncture. A randomized controlled design will be used with 144 children aged 7-12 years to be recruited between November 2024 and January 2025. Participants will be randomly assigned to control, sugared gum, or sugar-free gum groups. Pain and fear will be assessed using the Visual Analog Scale (VAS), Pen Pain Scale (PPS), and Children's Fear Scale (CFS). Crying duration will be recorded as a behavioral indicator. Data will be analyzed using Kruskal-Wallis, chi-square, and Spearman correlation tests with a significance level of p < .05. The study is intended to evaluate whether chewing gum can serve as a simple, low-cost, and non-invasive method to improve comfort and cooperation during pediatric venipuncture procedures.

DETAILED DESCRIPTION:
Needle-related procedures such as venipuncture are among the most common sources of pain, anxiety, and fear in pediatric clinical care. Negative experiences during these procedures may reduce cooperation, increase procedural difficulty, and contribute to long-term avoidance of healthcare settings. Identifying simple, low-cost, and non-pharmacological strategies to improve children's comfort during venipuncture is therefore an important clinical priority.

Chewing gum has been proposed as a potential method for modulating pain and anxiety through mechanisms such as distraction, rhythmic oral motor activity, and sensory engagement. Different gum types, including sugared and sugar-free varieties, may influence children's sensory experience differently. However, evidence regarding the use of chewing gum during pediatric procedures remains limited.

This randomized controlled study is designed to examine the effects of chewing sugared and sugar-free gum on pain, anxiety, and fear in children undergoing venipuncture. A total of 144 children aged 7-12 years will be recruited from outpatient clinical units between November 2024 and January 2025. Participants will be randomly assigned to one of three groups: a control group (no gum), a sugared gum group, or a sugar-free gum group. Children in the intervention groups will chew their assigned gum prior to and during venipuncture.

Pain will be measured using the Visual Analog Scale (VAS) and the Pen Pain Scale (PPS). Fear will be assessed using the Children's Fear Scale (CFS). Crying duration will be recorded as a behavioral indicator of distress. Demographic and clinical variables will also be collected to control for potential confounders.

Data will be analyzed using appropriate non-parametric and categorical statistical tests, including the Kruskal-Wallis test, chi-square test, and Spearman correlation analysis, with a predefined significance level of p < .05. The findings of this study are expected to contribute to the growing body of literature on non-pharmacological interventions for pediatric procedural support and may provide evidence for the integration of chewing gum as a practical technique to improve children's comfort and cooperation during venipuncture.

ELIGIBILITY:
Inclusion Criteria

* Children between 7-12 years of age
* Children requiring venous blood sampling
* Children able to chew gum safely
* Children who provide assent, with parental, legal guardian consent

Exclusion Criteria:

* Children with fever
* Children experiencing acute pain at the time of assessment
* Children who used analgesic medication within the previous four hours
* Children with medical conditions contraindicating gum chewing (e.g., jaw disorders)
* Children with allergy to gum ingredients
* Children with communication difficulties related to neurodevelopmental, hearing, visual impairments
* Children currently taking analgesic, sedative medications before the procedure

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Procedural Pain - Visual Analog Scale (VAS) | Immediately following the blood collection procedure (within a few minutes)
  Pain will be assessed using the Visual Analog Scale (VAS) to measure the severity of procedural pain during venipuncture in children assigned to control, sugared gum, or sugar-free gum groups. Units on a Scale. Minimum-Maximum Value: (0-10). Higher scores indicate worse pain
Procedural Pain - Pen Pain Scale (PPS) | Immediately following the blood collection procedure (within a few minutes)
  Pain will be assessed using the Pen Pain Scale (PPS) to measure the severity of procedural pain during venipuncture in children assigned to control, sugared gum, or sugar-free gum groups. Units on a Scale. Minimum-Maximum Value: (0-5): Higher scores indicate worse pain.
Procedural Fear - Children's Fear Scale (CFS) | Immediately following the blood collection procedure (within a few minutes)
  Fear will be assessed using the Children's Fear Scale (CFS) to measure the level of fear experienced by children during venipuncture in control, sugared gum, or sugar-free gum groups. Units on a Scale. Minimum-Maximum Value: (0-4). Higher scores indicate greater fear

SECONDARY OUTCOMES:
Duration of Crying During Venipuncture | From needle insertion until completion of venipuncture, with crying duration recorded in seconds, assessed for up to 5 minutes.
  Crying duration will be recorded as a behavioral indicator of distress in children during venipuncture in the control, sugared gum, and sugar-free gum groups.
Parent Satisfaction With Child's Blood Collection Experience | Immediately after completion of venipuncture (within 5 minutes).
  Parent satisfaction will be assessed as a Yes/No response to indicate whether the parent was satisfied with their child's experience during the blood collection procedure. Unit of Measure: Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Mus State Hospital, Pediatric Blood Collection Unit, Muş, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in de-identified form upon reasonable request to the Principal Investigator. Data will be available after publication of the main results and will be provided only for research purposes with appropriate ethical approval.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Sampallo Pedroza RM, Cardona Lopez LF, Ramirez Gomez KE. Description of oral-motor development from birth to six years of age. Rev Fac Med. 2015;62(4):593-604. Davas S, Kürtüncü M. The effect of three different methods during blood collection on pain level and parental satisfaction in children. Arch Health Sci Res. 2021;8(1):60-68. Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983;17(1):45-56. Beyaz E, Tüfekçi FG. Developing a new one-dimensional scale to measure pain in children: Pencil pain scale. J Pediatr Infants. 2021;4(1):1-10. McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: Preliminary investigation of the Children's Fear Scale. Health Psychol. 2011;30(6):780-788. Gülsoy H, Toru F, Öntürk Akyüz H, Üner FÖ. The impact of kaleidoscope and distraction cards on pain level during blood drawing in children. Med Res Rep. 2024;7(3):120-132.
- See also: Article on oral-motor development — https://doi.org/10.15446/revfacmed.v62n4.45211
- See also: Validation of VAS scale — https://doi.org/10.1016/0304-3959(83)90126-4
- See also: Distraction methods during pediatric blood draw — https://doi.org/10.55517/mrr.1408159
- See also: Distraction methods during pediatric blood draw — https://dergipark.org.tr/en/download/article-file/3613423